CLINICAL TRIAL: NCT04840134
Title: From Hardship to Hope: A Peer-led Intervention to Reduce Financial Hardship and Suicide Risk
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: In response to QA/compliance concerns about specific studies, NYSPI is undertaking an Institute-wide safety review of research protocols. Studies will resume recruitment after the review has confirmed they are deploying adequate safety protections.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: American Foundation for Suicide Prevention (Other); Baltic Street Wellness Solutions (Unknown)
Responsible Party: Principal Investigator, Oscar Jimenez-Solomon, PhD., MPH, Assistant Director, New York State Center of Excellence for Cultural Competence, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8078
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Suicide; Suicide Ideation; Suicidal Behavior; Hope; Financial Stress
MeSH Terms: conditions — Suicide; Financial Stress

STUDY DESIGN:
Intervention Model Description: This study evaluates the feasibility, acceptability, and initial efficacy of From Hardship to Hope (FHH) using a randomized controlled trial (RCT). The intervention arm will receive a 24-week peer-led financial wellness program in addition to clinical care with a licensed mental health clinician. The control arm will receive enhanced treatment as usual (eTAU), consisting of clinical care with a licensed mental health clinician plus information about financial wellness resources (a Financial Wellness Navigator and financial counseling handout).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- From Hardship to Hope: Financial Wellness Intervention (Experimental): Experimental: Participants in the experimental arm will receive "From Hardship to Hope, A Peer-led intervention to reduce financial hardship and suicide risk." The intervention will support individuals experiencing financial hardship and suicide risk to address their financial difficulties (e.g., debt, inability to meet basic needs) by coaching them on financial management techniques, facilitating a financial wellness plan, and connecting them with community-based financial supports (e.g., free financial counseling). The intervention will be facilitated by trained peer coaches, who are individuals with lived experience of financial hardship and suicidal ideation or suicidal behaviors who are state certified peer specialists (having met formal training and experience requirements).
  Interventions: Behavioral: From Hardship to Hope: A Peer-led intervention to reduce financial hardship and suicide risk
- Control Arm (Active Comparator): The control arm will receive enhanced treatment as usual (eTAU), consisting of clinical care with a licensed mental health clinician plus information about financial wellness resources (a Financial Wellness Navigator and financial counseling handout). The Financial Wellness Navigator is a curated document providing information about financial wellness resources available to New Yorkers (e.g., brief description of the service, eligibility criteria, website for more information, contact information). This directory will be provided via email, online link, and/or post mail, depending on participant preference.
  Interventions: Other: Enhanced Treatment as Usual (eTAU)

INTERVENTIONS:
Behavioral: From Hardship to Hope: A Peer-led intervention to reduce financial hardship and suicide risk — The intervention will be delivered in three consecutive phases:
  1. Intensive Intervention Phase (weeks 1 to 6), consisting of 6 weekly group sessions and 4 one-on-one coaching sessions to navigate financial resources.
  2. Intermediate Phase (weeks 7 to 12), consisting of 3 biweekly group sessions, and either 3 biweekly or 2 monthly one-on-one coaching sessions, based on participant preference.
  3. Follow up Phase (weeks 13 to 24), consisting of 3 monthly group sessions, and either 3 monthly or 6 biweekly one-on-one coaching sessions based on participant preference.
  Key intervention components:
  1. Peer-led group sessions
  2. Individual peer coaching sessions to complement group sessions
  Arms: From Hardship to Hope: Financial Wellness Intervention
Other: Enhanced Treatment as Usual (eTAU) — Enhanced Treatment as Usual (eTAU) consists of ongoing clinical care with a licensed mental health clinician, representing the current standard of care, plus provision of financial wellness informational resources. These resources include a Financial Wellness Navigator (a curated directory of financial wellness services available to New Yorkers) and a handout describing free financial counseling services and how to access them. The control condition does not include peer-led group sessions, individualized peer coaching, or warm referrals that are part of the From Hardship to Hope intervention.
  Arms: Control Arm

SUMMARY:
Financial hardship is an important risk factor for suicide. However, there are no evidence-based interventions to help individuals at risk for suicide to improve their financial situation. The intervention will support participants to address their financial difficulties (e.g., indebtedness, inability to meet basic needs) by coaching them to develop key financial management skills (e.g., budgeting, debt management), create a financial wellness action plan, map and activate their social networks, and connecting them with community-based financial supports (e.g., free financial counseling, publicly funded housing and food supports).

The intervention will be facilitated by trained peer coaches. The intervention will consist of three phases: (1) intensive; (2) intermediate; and (3) follow-up. The 6-week intensive phase will consist of 6 weekly group sessions and 4 one-on-one coaching sessions to navigate financial resources. The intermediate phase will consist of 3 biweekly group sessions, and either 3 biweekly or 2 monthly one-on-one coaching sessions, based on participant preference. The follow-up phase will offer 3 monthly group sessions, and either 3 monthly or 6 biweekly one-on-one coaching sessions based on participant preference. Group and one-on-one coaching sessions will be conducted remotely via a HIPAA-compliant videoconferencing platform.

This study will consist of five steps: (1) obtaining input from stakeholders to develop the intervention; (2) piloting it with a small sample of participants (n=10); (3) using this information to revise the intervention; (4) testing it in a randomized controlled trial with individuals experiencing financial hardship and suicide risk (n=96); and (5) finalizing the intervention manual.

DETAILED DESCRIPTION:
Decades of research have shown that financial hardship is a key risk factor for suicide. Studies have consistently found higher prevalence of suicidal ideation, suicide attempts, and suicide death among individuals experiencing financial hardship, such as unmanageable debts and difficulty paying for basic needs (e.g., housing, food). Stressful financial events (e.g., loss of income, evictions) are well-documented reasons for and precipitants of suicidal behavior. An increase in suicidal behavior is not only associated with objective aspects of financial hardship (e.g., number of debts, income level), but also with how hardship is experienced by individuals (e.g., financial threat, financial shame). In fact, growing evidence suggests that subjective financial hardship mediates the relationship between objective financial hardship and suicidal behavior.

Despite overwhelming evidence about the economic determinants of suicide, evidence-based interventions to reduce suicide risk and financial hardship are unavailable. Suicide prevention interventions at the individual level have largely focused on identifying or treating symptoms of psychiatric distress and other immediate clinical factors. Ecological-level interventions have mostly focused on increasing suicide awareness and reducing access to the means of suicide.

To address this gap, our project aims to develop a peer-led intervention that includes strategies and tools to reduce objective and subjective financial hardship, with the goal of decreasing hopelessness, shame, and depression (risk factors for suicide), increasing hope and life satisfaction (protective factors for suicide), and thereby reducing suicidal ideation and behaviors.

The main outcome of this study will be a manualized intervention to lessen financial hardship as a risk factor for suicidal ideation and behavior. If the findings of this study support its feasibility, acceptability, satisfaction, and initial efficacy, the investigators will formalize a peer coach training program, further develop an intervention fidelity measure, and pursue a randomized controlled trial to test intervention efficacy.

Specific aims and hypotheses are as follows:

1. With multi-stakeholder input, develop and iteratively revise From Hardship to Hope, a peer-led financial empowerment intervention with group and individual components to reduce SI/behaviors and financial hardship.
2. Assess the feasibility, acceptability, and satisfaction of the intervention using qualitative and quantitative methods.
3. Examine its initial efficacy by regular evaluations over 24 weeks on suicidal ideation (SI) severity and intensity, objective and subjective financial hardship, protective factors of suicide (e.g., hope, life satisfaction), and risk factors of suicide (e.g., hopelessness, depression). We hypothesize that, compared to the control arm, the intervention arm will show greater reductions in SI severity and intensity, hopelessness, and objective and subjective financial hardship, and greater increases in financial self-efficacy and hope from baseline to 24 weeks.
4. Explore the intervention's mechanisms of action (e.g., level of participation, subjective financial hardship). We hypothesize that the amount of change in SI severity and intensity will be positively correlated with the change in subjective financial hardship, and both will be associated with the level of participation.

ELIGIBILITY:
Inclusion Criteria:

* Working age (Self-reported age between 18-64).
* Provides informed consent (Self report: individual signs and dates Informed Consent Form).
* Stated willingness to comply with all study procedures and availability for the duration of the study (Self report).
* Lives or works in NYC (Self-report).
* Willing to receive referral to financial counseling (Self report).
* Objective financial hardship (Reports one or more types of financial hardship on the Financial Wellness Tool (FwTool), an 11-item assessment that measures overall financial hardship, food insecurity, housing hardship, difficulty paying for utilities, medical hardship, and indebtedness).
* Subjective financial hardship (Reports a Financial Threat score of 13 or higher [5-25] on the Financial Threat Scale (FTS), five-item scale that measures worry, fear, uncertainty, and preoccupation about one's financial situation).
* Moderate-to-high suicide risk as measured by the Columbia-Suicide Severity Rating Scale (C- SSRS) Screener administered by trained research staff (Endorses active suicidal ideation with or without a method or with some intent (items 2, 3, 4 on the C-SSRS) in the past 3 months, OR suicidal ideation with a plan or suicidal behavior (5 or 6 on the C-SSRS) in the past 3 months but NOT in the past month, confirmed by the study clinician during psychiatric evaluation).
* Receiving clinical treatment (Self-reports as currently enrolled in therapy or otherwise receiving treatment from a licensed mental health clinician; alternatively, willing to begin mental health treatment prior to the start of the intervention. Study participants will be asked to provide the name, phone number and email address for the treating clinician).
* Willing to participate in a financial wellness intervention via HIPAA-compliant videoconference platform (Self-report).
* Internet connection and video-capable device to participate in group sessions via HIPAA-compliant videoconference platform (Self-report).

Exclusion Criteria:

* Active SI with plan and intent in the past month (C-SSRS Screener administered by research staff and confirmed by study clinician (Yes to item 5, i.e., active suicidal ideation with plan and intent in the past month)).
* Recent suicidal behavior within the past month (C-SSRS Screener administered by research staff and confirmed by study clinician (Yes to item 6, i.e., has engaged in suicidal behaviors in the past month)).
* Florid psychosis or acute intoxication in need of detoxification (Clinical assessment by licensed study clinician during clinical evaluation).
* Cognitive impairment for those over age 60 (Montreal Cognitive Assessment - Blind Version (MoCA) conducted by research staff for those over age 60. (MoCA score below 19)).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
TFA: Theoretical Framework of Acceptability (TFA) Questionnaire Change | Week 1, Week 6, Week 12, Week 24
  A questionnaire designed to assess the acceptability of healthcare interventions across design, evaluation, and implementation phases. It consists of seven domains: affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy. The measure includes items assessing both prospective and retrospective acceptability.
TEI-SF: Treatment Evaluation Inventory Change | Week 1, Week 6, Week 12, Week 24
  A 9-item version of the original 15-item Treatment Evaluation Inventory, assessing treatment acceptability and ethical concerns.

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale - Intensity of Ideation Sub-scale Change | Baseline, Week 6, Week 12, Week 18, Week 24
  Interview-based assessment of suicide ideation intensity. It consists of 5 items measuring frequency, duration, controllability, deterrents, and reasons for Ideation. Sub-scale values range from 2 to 25. Higher scores indicate greater suicidal ideation intensity.
Beck Scale for Suicidal Ideation Change | Baseline, Week 6, Week 12, Week 18, Week 24
  21-item instrument for detecting and measuring the current intensity of specific attitudes, behaviors, and plans to die by suicide during the past week. The first 19 items assess the intensity of suicidality on a 3-point scale. Total score for these items ranges from 0 to 38, with greater scores indicating more severe suicidal ideation intensity. The final two items assess the number of previous suicide attempts and the severity of the intent to die associated with the last attempt.
Economic Hardship Questionnaire Change | Baseline, Week 6, Week 12, Week 18, Week 24
  12-item self-report scale measuring family economic hardship and changes in a household's style of living in the past 6 months (e.g., drop in income, ability meet basic needs). Values range from 0 to 36. Higher scores indicate greater recent economic hardship.
E-FwT: ENGAGE Financial Wellness Tool Change | Baseline, Week 6, Week 12, Week 18, Week 24
InCharge Financial Distress/Financial Well-Being Scale (IFDFW) Change | Baseline, Week 6, Week 12, Week 18, Week 24
  An 8-item self-report scale assessing financial distress and well-being on a continuum. Higher scores indicate greater financial well-being, while lower scores reflect higher financial distress. The scale provides a subjective measure of an individual's financial situation based on perceived stress and stability.
Financial Hardship Screener | Baseline, Week 6, Week 12, Week 18, Week 24

OTHER OUTCOMES:
Financial Satisfaction Scale | Baseline, Week 6, Week 12, Week 18, Week 24
Financial Threat Scale Change | Baseline, Week 6, Week 12, Week 18, Week 24
  5-item self-report measure of current feelings of worry and preoccupation with current financial situation. Scores range from 5 to 25. Greater scores indicate higher perceived financial threat.
Satisfaction with Life Scale Change | Baseline, Week 6, Week 12, Week 18, Week 24
  5-item self-report measure of global current life satisfaction. Values range from 5 to 35. Higher scores indicate greater levels of life satisfaction.
Medical Outcomes Survey Social Support Scale (MOS-SSS) Change | Baseline, Week 6, Week 12, Week 18, Week 24
  19-item measure of perceived current social support in emotional/informational, tangible, affectionate, and positive social interactions. Values range from 0 to 100. Higher scores indicate greater social support.
UCLA Loneliness Scale-8 (ULS-8) Change | Baseline, Week 6, Week 12, Week 18, Week 24
  8-item measure of perceived social isolation. Values range from 8 to 32. Higher scores indicate higher levels of loneliness.
State Shame and Guilt Scale (SSGS) | Baseline, Week 6, Week 12, Week 18, Week 24
  The SSGS is a self-rating scale of in-the-moment (state) feelings of shame, and guilt experiences. Ten items (five for each of the two subscales) are rated on a 5-point scale Likert scale.
Beck Hopelessness Scale Change | Baseline, Week 6, Week 12, Week 18, Week 24
  20-item self-report measure of hopelessness about the future, loss of motivation, and poor expectations in the past week. Values range from 0 to 20. Higher scores indicate higher levels of hopelessness.
E-SF: The Entrapment Scale Short-Form | Baseline, Week 6, Week 12, Week 18, Week 24
  A shortened version of the 16-item Entrapment Scale, measuring feelings of being trapped in distressing situations. Designed for individuals at elevated suicide risk, with higher scores indicating greater perceived entrapment.
Patient Health Questionnaire (PHQ-9) Change | Baseline, Week 6, Week 12, Week 18, Week 24
  9-item measure of depressive symptoms and severity in the past two weeks. Values range from 0 to 27. Higher scores indicate greater depression severity.
GAD-7: Generalized Anxiety Disorder 7-item | Baseline, Week 6, Week 12, Week 18, Week 24
  The Generalized Anxiety Disorder 7 Item Scale (GAD-7) is a brief self-report questionnaire designed to screen for and measure the severity of generalized anxiety disorder. The GAD-7 consists of seven questions that assess the frequency of anxiety symptoms over the past two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Jimenez-Solomon, PhD, MPH, Principal Investigator — New York State Psychiatric Institute, Columbia University Irving Medical Center
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No